CLINICAL TRIAL: NCT03965845
Title: A Phase 1b/2, Open Label, Dose Escalation and Expansion Study of the Glutaminase Inhibitor Telaglenastat (CB-839) in Combination With CDK4/6 Inhibitor Palbociclib in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of Telaglenastat (CB-839) in Combination With Palbociclib in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-012
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumors; NSCLC; CRC; KRAS Gene Mutation
Keywords: Tumor Metabolism; Glutaminase Inhibitor; CB-839; Palbociclib; PALBO; Telaglenestat; CDK4/6; CDK4; CDK6
MeSH Terms: interventions — CB-839; palbociclib; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Telaglenastat 600 mg and Palbociclib 75 mg (Experimental)
  Interventions: Drug: Telaglenestat (CB-839); Drug: Palbociclib Oral Capsule or Tablet [Ibrance]
- Cohort 2: Telaglenastat 800 mg and Palbociclib 75 mg (Experimental)
  Interventions: Drug: Telaglenestat (CB-839); Drug: Palbociclib Oral Capsule or Tablet [Ibrance]
- Cohort 3: Telaglenastat 800 mg and Palbociclib 100 mg (Experimental)
  Interventions: Drug: Telaglenestat (CB-839); Drug: Palbociclib Oral Capsule or Tablet [Ibrance]
- Cohort 3: Telaglenastat 800 mg and Palbociclib 125 mg (Experimental)
  Interventions: Drug: Telaglenestat (CB-839); Drug: Palbociclib Oral Capsule or Tablet [Ibrance]
- Part 2: Expansion (Experimental): The recommended phase 2 dose (RP2D) determined from Part 1 will be the treatment for all cohorts in expansion Part 2.
  Interventions: Drug: Telaglenestat (CB-839); Drug: Palbociclib Oral Capsule or Tablet [Ibrance]

INTERVENTIONS:
Drug: Telaglenestat (CB-839) — Teleglenastat is an oral tablet administered twice daily with food at the assigned dose level. Dose is taken with palbociclib each day in 28-day cycles.
Drug: Palbociclib Oral Capsule or Tablet [Ibrance] — Palbociclib (Ibrance) is an oral capsule or tablet administered once daily with food on Days 1-21 of every 28-day cycle in combination with telaglenestat. Days 22-28 of every cycle, palbociclib is not taken.
  Other Names: Ibrance

SUMMARY:
This is a Phase 1b/2 study to determine the recommended phase 2 dose (RP2D), safety and tolerability, pharmacokinetics (PK) and clinical activity of the glutaminase inhibitor telaglenestat (CB-839) with the CDK4/6 Inhibitor, palbociclib in participants with advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Have documented incurable/locally advanced or metastatic solid tumors that have either relapsed or are refractory or intolerant to the standard therapies of proven clinical benefit.
* Part 2: Availability of archival tumor tissue block or slides (Fresh tumor biopsy will be required if archival tissue is not available)
* Part 2, Cohort 1: Incurable/locally advanced or metastatic KRAS-mutant CRC previously treated with systemic therapy (examples include: oxaliplatin-, irinotecan-and 5 FU-based chemotherapy (unless contraindicated) with or without bevacizumab)
* Part 2, Cohort 2: Incurable/locally advanced or metastatic KRAS-mutant NSCLC previously treated with systemic chemotherapy including platinum-based and anti-PD-1/PDL-1 therapy (unless contraindicated)
* Part 2, Cohort 3: Advance KRAS-mutant Pancreatic Ductal Adenocarcinoma (PDAC) harboring a mutation or loss in CDKN2A (PDAC) and received treatment with one or more lines of systemic chemotherapy with FOLFIRINOX and/or gemcitabine/abraxane in the neoadjuvant, adjuvant, or metastatic disease setting or unable to receive standard of care chemotherapy

Cohort 4 may be opened only if Cohort 3 achieves predefined criteria for efficacy

-Part 2 Cohort 4: Advanced KRAS-mutant Pancreatic Ductal Adenocarcinoma (PDAC). · Histological or cytological diagnosis of advanced or metastatic KRAS-mutant with CDKN2A wild type (PDAC) and received treatment with one or more lines of systemic chemotherapy with FOLFIRINOX and/or gemcitabine/abraxane in the neoadjuvant, adjuvant, or metastatic disease setting or unable to receive standard of care chemotherapy.

For both Part 1 and 2:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Ability to provide written consent in accordance with federal, local and institutional guidelines
* PER RECIST v1.1 evaluable disease (for part 1) or measurable disease (for Part 2)
* Recovery to baseline or to Grade 1 CTCAE v5.0 of toxicities that were related to prior therapies

Exclusion Criteria:

* Prior treatment with CB-839 or palbociclib
* Unable to receive oral medication
* Infection requiring more than 5 days of parenteral antibiotics, antivirals, or antifungals within two weeks prior to C1D1
* Unable to discontinue proton pump inhibitor use before study treatment
* Refractory nausea and vomiting, uncontrolled diarrhea, malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes or other situation that may preclude adequate absorption
* Active and/or untreated central nervous system metastasis. Patients with treated brain metastasis must have (1) documented radiographic stability of at least 4 weeks in duration demonstrating on baseline central nervous system imaging prior to study treatment and (2) be symptomatically stable and off steroids for at least 2 weeks before administration of any study treatment.
* Major surgery within 28 days prior to first dose of study drug
* Receipt of any anticancer therapy within the following windows:

  1. small molecule TKI therapy (including investigational) within 2 weeks or 5 half-lives prior to expected Cycle 1 Day 1 dose
  2. any type of anti-cancer antibody or cytotoxic chemo within 4 weeks prior to Cycle 1 Day 1 Dose
  3. radiation therapy for bone metastasis within 2 weeks prior or any other external radiation therapy within 4 weeks prior to C1D1
  4. patients with clinically relevant ongoing complications from prior radiation therapy are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of telaglenestat (CB-839) in combination with palbociclib: (CR) number of participants with treatment related adverse events | Start of treatment to 28 days post treatment
  Number of participants with treatment related adverse events as assessed by CTCAE v5.0
Maximum tolerated dose and/or Recommended Phase 2 Dose: | Measured from Part 1 patients only within their first 28 day cycle
  Incidence and nature of dose-limiting toxicities

SECONDARY OUTCOMES:
Maximum plasma concentration of telaglenastat and palbociclib: | PKs are drawn on two different days (Day 8 and Day 15) during Cycle 1
  Non-compartmental method of analysis will be used to analyze the plasma concentrations
Anti-tumor activity of telaglenestat and palbociclib: | Approximately every 8 weeks until disease progression, for approximately 18 months
  Change in tumor size from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emil Kuriakose, MD, Study Director — Calithera Biosciences, Inc
Locations (10):
- United States (10):
  - UCLA Hematology/Oncology, Santa Monica, California
  - Emory, Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Regions Cancer care Center, Saint Paul, Minnesota
  - Sarah Cannon Research Institute- Tennessee Oncology, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - South Texas Accelerated Research Therapeutic, LLC, San Antonio, Texas
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No